CLINICAL TRIAL: NCT07326384
Title: Assessment of Psychiatric Problems in Pre- and Post-Intervention in Patients With Congenital Heart Disease: A Prospective Cohort Study.
Brief Title: Assessment of Psychiatric Problems in Pre- and Post-Intervention in Patients With CHD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shrouk Alaa-eldein Abdallah, Cardiology resident at Assiut University Heart Hospital, Assiut University
Other Study IDs: Interventions in CHD
Record Dates: First submitted 2025-09-30; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; Psychiatric problems; Mental health and cardiovascular disease; Cardiac intervention
MeSH Terms: conditions — Heart Defects, Congenital; Psychological Well-Being; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult
  Interventions: Procedure: Cardiac interventions
- Child
  Interventions: Procedure: Cardiac interventions

INTERVENTIONS:
Procedure: Cardiac interventions — surgical or catheter-based, Corrective or palliative.

SUMMARY:
The goal of this observational study is to learn about the relationship between cardiac intervention and subsequent psychiatric symptoms in patients with CHD. Due to the known high prevalence of mental health issues-with up to 50% of adults and 35% of pediatric patients with CHD experiencing mood or anxiety disorders-this research is crucial for improving long-term psychosocial care.

The main questions it aims to answer are:

* What is the prevalence of psychiatric problems in CHD patients?
* Do psychiatric problems change or evolve after a cardiac intervention?
* Who Can Take Part (Supporting Information)

The study is actively recruiting patients who meet specific criteria:

* Diagnosed with CHD and scheduled for a palliative or corrective cardiac intervention (surgical or catheter-based).
* Patients of both genders can participate.

Patients cannot take part if they have:

* A current or pre-existing psychiatric or neurological disorder. - How the Research Will Happen

This is a prospective, longitudinal cohort study that tracks the same participants over time. Participants will be asked to complete a series of validated psychological and cognitive assessments at three specific time points:

* T0 (Baseline): Before the cardiac procedure.
* T1 (Short-term): Approximately 1 month after the procedure.
* T2 (Long-term): Approximately 3 months after the procedure.

Participants will complete standardized measures covering a wide range of topics, including:

* Psychological symptoms (e.g., depression, anxiety).
* Cognitive function (e.g., memory and attention).
* Sleep quality.
* Eating attitudes.
* Suicidal ideation. Potential Benefits: This research is critical for identifying dynamic changes in mental health related to cardiac procedures and will help the medical community understand the psychological impact of these interventions, leading to better screening and long-term quality of life.

ELIGIBILITY:
1. Inclusion criteria:

   * patients of both gender.
   * Confirmed diagnosis of congenital heart disease requiring surgical or catheter-based intervention.
2. Exclusion criteria:

   * current or a pre-existing psychiatric or neurological disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with congenital heart disease presenting for palliative or corrective cardiac intervention (surgical or catheter-based).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of psychiatric disorders in adults with congenital heart disease, as assessed by the Symptom Checklist-90-Revised (SCL-90-R) Global Severity Index. | At baseline, Pre-procedure visit (within 4 weeks of intervention).
  * Measurement Tool: Symptom Checklist-90-Revised (SCL-90-R).
  * Unit of Measure: Units on a Scale (Global Severity Index T-score).
Prevalence of psychiatric disorders in children with congenital heart disease, as assessed by the Child Behavior Checklist (CBCL) Total Problems T-score. | At baseline, pre-procedure visit (within 4 weeks of intervention).
  * Measurement Tool: Child Behavior Checklist (CBCL).
  * Unit of Measure: Units on a Scale (Total Problems T-score).